CLINICAL TRIAL: NCT00848666
Title: Safety and Efficacy of a Novel Topical Therapy for Tinea Pedis (Athlete's Foot)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Michael Kahana, Hillel Yaffe Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC 48-08
Record Dates: First submitted 2008-08-28; First posted 2009-02-20 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Patients with tinea pedis
  Interventions: Drug: Topical therapy

INTERVENTIONS:
Drug: Topical therapy — One time immersion of the feet in a liquid containing water, alcohol, vinegar, benzoic acid and salicylic acid for a total of 30 minutes.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a novel topical therapy in patients with laboratory confirmed tinea pedis. During the follow-up period clinical and mycological examinations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy patients with laboratory proven tinea pedis

Exclusion Criteria:

* Age lower than 18 and higher than 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Cure of tinea pedis | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel